CLINICAL TRIAL: NCT04626453
Title: Muscular and Cerebral Oxygenation Changes After Moderate-Intensity Exercise in Sedentary Older Adults With Type 2 Diabetes
Brief Title: Oxygenation Changes After 2-month Exercise in Sedentary Older Adults With Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Fei Zhao, Ph.D. candidate student, MPT, State University of New York at Buffalo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00004297
Record Dates: First submitted 2020-10-30; First posted 2020-11-12 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Diabetes Mellitus, Type 2; Oxygen Deficiency
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypoxia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- sedentary older adults with Type 2 Diabetes (Experimental): Sedentary older adults with Type 2 Diabetes as the intervention group will do a 2-month home exercise.
  Interventions: Behavioral: 2-month home moderate-intensity exercise
- Active older adults with Type 2 Diabetes (No Intervention): Active older adults with Type 2 Diabetes will not do exercise.
- Healthy older adults (No Intervention): Healthy older adults will not do exercise.

INTERVENTIONS:
Behavioral: 2-month home moderate-intensity exercise — The 2-month exercise will be conducted at the participants' homes. Participants will be recommended to perform the combined exercise, which consists of the resistance exercise and walking at a faster speed than leisure walking at a moderate-intensity, for 6 days/week. They can decide which day they won't perform the exercise. Participants will be encouraged to do progressive resistance exercise and walking twice a day, once in the morning and the other time in the afternoon. Resistance exercise will be suggested to perform every other day for three days/week and walking as the aerobic exercise will be on alternate days for three days/week.
  Arms: sedentary older adults with Type 2 Diabetes

SUMMARY:
The aim of the study is to determine the physiological evidence of how muscular and cerebral oxygenation changes link to fatigue, physical, and cognitive performance after moderate-intensity exercise in sedentary older adults with type 2 diabetes.

DETAILED DESCRIPTION:
This is an experimental design. One intervention group will do exercise for 2 months and be measured twice, at baseline, and after 2 months. The other 2 control groups will be assessed just once without exercise intervention. Our primary objective is to clarify physiological evidence of how muscular and cerebral oxygenation changes in sedentary older adults with diabetes after low-to-moderate intensity exercise. The secondary objective is to determine fatigue, physical, cognitive performance changes, blood glucose level among sedentary older adults with diabetes after low-to-moderate intensity exercise.

ELIGIBILITY:
Inclusion Criteria:

* For the intervention group, the inclusion criteria are

  * sedentary older adults 60 years or older who are living in their homes in the community
  * diagnosed type 2 diabetes
  * ambulatory with or without mobility devices such as a cane and/or walker
  * Be able to follow simple exercise instructions without assistance.
* For the comparison group, the inclusion criteria are

  * individuals aged 60 years or older who are living in their homes, in the community;
  * ambulatory with or without devices;
  * able to follow simple exercise instructions without assistance
  * able to walk six minutes as quickly as possible without any adverse symptoms including extreme pain on feet or joints, dizziness, vertigo, or nausea.

Exclusion Criteria:

* For the intervention group, the exclusion criteria are

  * foot deformities, cuts, blisters, or amputation, Achilles tendonitis, joint replacements within the past three months, Parkinson's disease, retinopathy such as severe glaucoma, current or uncontrolled vestibular disorders
  * current smoking or smoking within the last 12 months
  * current cardiopulmonary diseases, vascular disease, or stroke
  * dementia indicating the inability to follow exercise instructions independently
  * those who are currently or plan to receive physical therapy in the following three months
  * individuals without English proficiency will be excluded
  * If the individuals with blood glucose level are over 400 mg/dL or HbA1C > 8.0%, and
  * type 1 diabetes.

For the comparison group, the exclusion criteria are

* individuals who have prediabetes, diabetes, or current cardiopulmonary diseases and stroke
* current smoking or smoking within the last 12 months
* individuals with foot deformities, cuts, blisters, or amputation, Achilles tendonitis, joint replacements within the past three months, Parkinson's disease, retinopathy such as severe glaucoma, current or uncontrolled vestibular disorders, and dementia.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2020-10-29 (Actual); Primary Completion 2021-06-27 (Actual); Study Completion 2021-06-27 (Actual)

PRIMARY OUTCOMES:
normalized ∆SmO2 rate | measure twice, at baseline and after 2 months
  a parameter of muscular oxygenation to indicate the match or mismatch between oxygen supply and oxygen demand during the physical stimulus.
recovery time | measure twice, at baseline and after 2 months
  a parameter of muscular oxygenation, time taken in seconds after the exercise to back to the beginning oxygenation level.
Resting SmO2 | measure twice, at baseline and after 2 months
  a parameter of muscular oxygenation, the average oxygenation level in % while sitting still for 3 minutes before doing physical performance tests.
Oxyhemoglobin differences | measure twice, at baseline and after 2 months
  a parameter of cerebral oxygenation, the difference of the oxyhemoglobin in mL per gram before and after the cognitive tests.

SECONDARY OUTCOMES:
Fatigue | measure twice, at baseline and after 2 months
  Fatigue will be assessed by the Numeric Fatigue Scale (NFS) by selecting a number from 0 to 10. 0 is no fatigued at all, 10 is extremely fatigued.
Timed Up and Go test score in seconds | measure twice, at baseline and after 2 months
  An assessment of physical performance. Time in seconds from sitting up from a chair, walking to 3 meters, turning, walking back to sitting down on a chair.
Short Physical Performance Battery | measure twice, at baseline and after 2 months
  An assessment of physical performance. This test contains three sections: balance, walking speed and chair stand. The scores are 0-12.
Bilateral Heel Raise test | measure twice, at baseline and after 2 months
  An assessment of physical performance. This test askes to do heel raise to the maximum height continuously. Time to fatigued in seconds and the frequencies of heel raise are recorded.
6 Minute Walking Test | measure twice, at baseline and after 2 months
  An assessment of physical performance. The test assesses time in seconds when participants walk as fast as they can in 6 minutes.
Mini-cog test | measure twice, at baseline and after 2 months
  An assessment of cognitive performance. A Short term memory test.
Trail Making Test | measure twice, at baseline and after 2 months
  An assessment of cognitive performance. A executive function test.
blood glucose level in mg/dL | measure twice, at baseline and after 2 months
  Blood glucose level before and after exercise

CONTACTS AND LOCATIONS:
Overall Officials: Fei Zhao, Principal Investigator — University at Buffalo
Locations (1):
- University at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No